CLINICAL TRIAL: NCT01112631
Title: Prospective Comparison of Quality of Life and Cardiopulmonary Morbidity After Surgery in Non-small Cell Lung Cancer Patients Treated With and Without Postoperative Radiotherapy
Brief Title: Prospective Study of Quality of Life in Non-small Cell Lung Cancer (NSCLC) Patients Treated With/Without Postoperative Radiotherapy
Status: Completed | Type: Observational
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: Institute of Tuberculosis and Lung Diseases in Warsaw (Unknown); The Greater Poland Centre of Lung Diseases and Tuberculosis in Poznan (Unknown); The Greater Poland Cancer Centre (Other); Cancer Centre in Bydgoszcz (Unknown); Kujawsko-Pomorskie Center of Pulmonology in Bydgoszcz (Unknown); Specialized Hospital in Zdunowo - Szczecin (Unknown); Regional Cancer Hospital - Szczecin (Unknown); Medical University of Gdansk (Other); Holycross Cancer Center in Kielce (Unknown); Department of Thoracic Surgery - Wrocław (Unknown); Department of Radiotherapy - Olsztyn (Unknown); Department of Thoracic Surgery - Łódź (Unknown); Lower Silesian Oncology Center - Wroclaw (Unknown); Regional Specialized Hospital -Chęciny, Czerwona Góra (Unknown); Department of Thoracic Surgery - Otwock (Unknown); Medical University of Łódź (Other)
Responsible Party: Prof Krzysztof Bujko, Maria Sklodowska-Curie Memorial Cancer Center, Institute of Oncology in Warsaw
Other Study IDs: LPSG01
Record Dates: First submitted 2010-04-27; First posted 2010-04-28 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2010-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC,; PORT,; Quality of Life,; Pulmonary function after RT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Stage II patients post surgery: Stage II patients treated with surgery alone
- Stage III patients post surgery: Stage III patients treated with surgery and PORT

SUMMARY:
The patients from 12 centers were included into the study. pN2 patients received PORT, pN1 patients did not. PORT was 3D-planned and consisted in 54-56 Gy in 27-28 fractions. One month after surgery, all patients completed EORTC QLQ C-30 questionnaires and had pulmonary function tests (PFT); cardiopulmonary symptoms were assessed by modified LENT-SOM score. Two years after, all patients free of disease repeated the same examinations. Changes in QLQ, LENT-SOM score and the results of PFT were compared for patients receiving and not PORT.

ELIGIBILITY:
Inclusion Criteria:

* complete resection by lobectomy, bi-lobectomy or pneumonectomy of NSCLC,
* pN1 or pN2 disease,
* signed informed consent for participation in the study,
* Karnofsky Performance Status (KPS) higher than 70%.

Exclusion Criteria:

* presence of distant metastases,
* N2 diagnosed before surgery in imaging and/or mediastinoscopy,
* previous radiotherapy to the chest,
* no or inadequate mediastinal nodal dissection ,
* FEV1 after surgery lower than 1.0 liter,
* any active infectious process (including fistula formation) in the chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It was assessed that during planned 3 years of accrual approximately 360 stage II patients treated with surgery alone and approximately 240 stage III patients treated with surgery and postoperative radiotherapy (PORT) would enter the study.The higher number of inclusions of pN1 was planned, because of expected higher percentage of cancer related deaths within two years in pN2 patients.
  Patients with pN1 disease were followed in the thoracic surgery center and had no PORT. Patients with pN2 disease were referred to PORT.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2003-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | One month after surgery and two years after postoperative radiotherapy or surgery alone
  All patients had pulmonary function tests (PFT) with Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1) recorded.

SECONDARY OUTCOMES:
Quality of Life | One month after surgery and two years after postoperative radiotherapy or surgery alone
  For quality of life assessment, patients were asked to complete the Quality of Life Questionnaire Core 30 Items (QLC-C30) of the European Organization for Research and Treatment of Cancer (EORTC).

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bujko, Prof., Principal Investigator — Roentgena 5, 02-781 Warsaw, Poland
Locations (1):
- M. Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland

REFERENCES:
- [Background] Kepka L, Bujko K. [Postoperative radiotherapy for non-small cell lung cancer: evidence based data and clinical practice]. Pneumonol Alergol Pol. 2007;75(3):256-61. Polish. PMID 17966101